CLINICAL TRIAL: NCT05398926
Title: An Open Clinical Trial to Evaluate Immunogenicity and Safety of a Third Dose at Different Times After Two-dose of COVID-19 Vaccine (Vero Cell), Inactivated in the Elderly Aged 60 Years and Above
Brief Title: Immunogenicity and Safety of a Third Dose of COVID-19 Vaccine(Vero Cell), Inactivated in the Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-nCoV-4011
Record Dates: First submitted 2022-05-31; First posted 2022-06-01 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines; sinovac COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental group 1 (3-month interval) (Experimental): 100 subjects who have received two doses of COVID-19 vaccine (Vero cell), Inactivated will receive a 3rd dose of the vaccine (3-month interval）.
  Interventions: Biological: COVID-19 Vaccine (Vero cell), Inactivated
- Experimental group 2 (4-month interval) (Experimental): 100 subjects who have received two doses of COVID-19 vaccine (Vero cell), Inactivated will receive a 3rd dose of the vaccine (4-month interval）.
  Interventions: Biological: COVID-19 Vaccine (Vero cell), Inactivated
- Experimental group 3 (5-month interval) (Experimental): 100 subjects who have received two doses of COVID-19 vaccine (Vero cell), Inactivated will receive a 3rd dose of the vaccine (5-month interval）.
  Interventions: Biological: COVID-19 Vaccine (Vero cell), Inactivated
- Experimental group 4 (6-month interval) (Experimental): 100 subjects who have received two doses of COVID-19 vaccine (Vero cell), Inactivated will receive a 3rd dose of the vaccine (6-month interval）.
  Interventions: Biological: COVID-19 Vaccine (Vero cell), Inactivated

INTERVENTIONS:
Biological: COVID-19 Vaccine (Vero cell), Inactivated — The COVID-19 vaccine,inactivated was manufactured by Sinovac Research& Development Co., Ltd.600SU inactivated SARS-CoV-2 CZ strain virus in 0.5 mL of aluminium hydroxide solution per injection.
  Other Names: CoronaVac®

SUMMARY:
This is an open phase Ⅲ clinical trial of COVID-19 vaccine (Vero cell), inactivated manufactured by Sinovac Research & Development Co., Ltd.The purpose of this study is to evaluate Immunogenicity and safety of a third dose at different times after two-dose of COVID-19 vaccine (Vero cell), Inactivated in the Elderly Aged 60 years and above.

DETAILED DESCRIPTION:
This study is an open phase Ⅲ clinical trial. The main purpose of this study is to evaluate Immunogenicity and safety of a third dose at different times after two-dose of COVID-19 vaccine (Vero cell), Inactivated manufactured by Sinovac Research & Development Co., Ltd. in the elderly aged 60 years and above.A total of 400 subjects aged 60 years and above who had received two doses of COVID-19 vaccine(Vero Cell), inactivated manufactured by Sinovac Research & Development Co., Ltd. between 3 - 6 months ago (100 subjects for 3 months, 4 months, 5 months and 6 months,respectively) will be enrolled and receive a third dose of two-dose of COVID-19 vaccine (Vero cell), inactivated were enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 60 years and above;
* Provide legal identification;
* Have completed two-dose of COVID-19 vaccine (Vero cell), inactivated manufactured by Sinovac Research& Development Co., Ltd. for 3~6 months（The interval between two doses was 21~35 days）；
* Be able to understand and voluntarily sign the informed consent form and be willing to complete the study according to the research plan.

Exclusion Criteria:

* History of SARS-CoV-2 infection(laboratory confirmed);
* Those who have received COVID-19 vaccine from other manufacturers other than Sinovac Research& Development Co., Ltd., or who have received booster immunization with COVID-19 vaccine after two doses of COVID-19 vaccine (Vero cell),inactivated manufactured by Sinovac Research& Development Co., Ltd.;
* History of serious adverse reactions to the vaccine or vaccine components, such as urticaria dyspnea and angioneuroedema;
* Autoimmune disease or immunodeficiency/immunosuppression;
* Severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver or kidney diseases, malignant tumors, etc;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids(excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months or plan to receive these treatments during the study period;
* Receipt of blood products within in the past 3 months or plan to receive these treatments during the study period;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days,or receipt of inactivated or subunit vaccines in the past 7 days;
* Onset of various acute or chronic diseases within 7 days prior to the study;
* Axillary temperature >37.0°C;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 400 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Immunogenicity index-GMT of neutralizing antibodies | At 14 days after vaccination
  GMT of neutralizing antibodies at 14 days after vaccination
Immunogenicity index- GMT of neutralizing antibodies | At 28 days after vaccination
  GMT of neutralizing antibodies at 28 days after vaccination
Safety index-Incidence of adverse reactions | 0~28 days after vaccination
  Incidence of adverse reactions 0~28 days after vaccination

SECONDARY OUTCOMES:
Immunogenicity index-seropositive rate of neutralizing antibodies | Day 0 before vaccination and 14 days, 28 days and 180 days after vaccination
  Seropositive rate of neutralizing antibodies of neutralizing antibodies before vaccination and at different points after vaccination
Immunogenicity index-GMT of neutralizing antibodies | Day 0 before vaccination and 180 days after vaccination
  GMT of neutralizing antibodies before vaccination and at different points after vaccination.
Immunogenicity index-4-fold increase rate of neutralizing antibodies | At 14 days and 28 days after vaccination.
  4-fold increase rate of neutralizing antibodies at different points after vaccination.
Safety index-Incidence of adverse reactions | 0~7 days after vaccination
  Incidence of adverse reactions 0~7 days after vaccination.
Safety index-Incidence of serious adverse events | 6 months after vaccination
  Incidence of serious adverse events 6 months after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yang, Master, Principal Investigator — Yunnan Provincial Center for Disease Control and Prevention
Locations (1):
- Yongde Center for Diseases Control and Prevention, Lincang, Yunnan, China